CLINICAL TRIAL: NCT01612000
Title: Phase 2 Observer-Blind, Randomized Trial to Evaluate the Immunogenicity and Safety of PanBlok at Three Dose Levels Adjuvanted With a Stable Oil-in-Water Emulsion Compared With PanBlok Without Adjuvant in Healthy Adults Aged 18 to 49 Years
Brief Title: Safety and Immunogenicity of PanBlok Influenza Vaccine in Healthy Adults
Acronym: PSC25
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSC25
Record Dates: First submitted 2012-05-07; First posted 2012-06-05 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PanBlok 15µg in 2% SE (Experimental): 15µg recombinant hemagglutinin in a 2% oil-in-water stable emulsion (rHA adjuvant). 0.5mL intramuscular injection on Day 0 and Day 21 in the deltoid muscle
  Interventions: Biological: PanBlok; Biological: rHA adjuvant
- PanBlok 3.8µg in 2% SE (Experimental): 3.8µg recombinant hemagglutinin in a 2% oil-in-water stable emulsion (rHA adjuvant). 0.5mL intramuscular injection on Day 0 and Day 21 in the deltoid muscle
  Interventions: Biological: PanBlok; Biological: rHA adjuvant
- PanBlok 7.5µg No Adjuvant (Experimental): 7.5µg recombinant hemagglutinin, no adjuvant. 0.5mL intramuscular injection on Day 0 and Day 21 in the deltoid muscle
  Interventions: Biological: PanBlok
- PanBlok 7.5µg in 2% SE (Experimental): 7.5µg recombinant hemagglutinin in a 2% oil-in-water stable emulsion (rHA adjuvant). 0.5mL intramuscular injection on Day 0 and Day 21 in the deltoid muscle
  Interventions: Biological: PanBlok; Biological: rHA adjuvant

INTERVENTIONS:
Biological: PanBlok — Intramuscular injection
  Other Names: rHA; recombinant hemagglutinin
Biological: rHA adjuvant — Intramuscular injection
  Other Names: SE
  Arms: PanBlok 15µg in 2% SE; PanBlok 3.8µg in 2% SE; PanBlok 7.5µg in 2% SE

SUMMARY:
The purpose of this study is to investigate the safety and immunogenicity of a recombinant hemagglutinin (rHA) influenza vaccine derived from A/Indonesia/05/2005 (H5N1) administered at 3 dose levels in adjuvanted (SE) rHA formulations and 1 dose levels in an un-adjuvanted rHA formulation.

DETAILED DESCRIPTION:
All currently licensed influenza vaccines in the United States are produced in embryonated hen's eggs. There are several well-recognized disadvantages to the use of eggs as the substrate for influenza vaccine. Eggs require specialized manufacturing facilities and could be difficult to scale up rapidly in response to an emerging need such as a pandemic. It is usually necessary to adapt candidate vaccine viruses for high-yield growth in eggs, a process that can be time consuming, is not always successful, and can select receptor variants that may have suboptimal immunogenicity. In addition, agricultural diseases that affect chicken flocks, and that might be an important issue in a pandemic due to an avian influenza virus strain, could easily disrupt the supply of eggs for vaccine manufacturing. Therefore, development of alternative substrates for influenza vaccine production has been identified as a high-priority objective.

One potential alternative method for production of influenza vaccine is expression of the influenza virus hemagglutinin (HA) using recombinant DNA techniques. This alternative avoids dependence on eggs and is very efficient because of the high levels of protein expression under the control of the baculovirus polyhedrin promoter.

ELIGIBILITY:
Inclusion Criteria:

* Young adults aged 18-49 years
* Able to give written informed consent to participate.
* Vital signs within normal limits.
* The subject must be in good health as determined by targeted physical examination, when necessary, based on medical history. Stable medical condition is defined as: no recent change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company, etc., or is done for financial reasons, as long as in the same class of medication, will not be considered a violation of the inclusion criterion. Any change to prescription medication due to improvement of a disease outcome will not be considered a violation of the inclusion criterion.
* Comprehensive Metabolic Panel and other tests for the following must fall within normal limits or not exceed a Grade 1 abnormality at screening. Any Grade 1 abnormality must be clinically acceptable to the investigator in the context of other parameters such the subject's medical history. However, this will not apply to an above the upper limit of the normal range for ALT. Subjects with values above the upper limit of the normal range for ALT at the screening visit will not be enrolled.
* Complete Blood Count with Cell Differential and urinalysis must fall within normal limits at screening except when clinically acceptable to the investigator in the context of other parameters such the subject's medical history.
* Women of child-bearing potential (WOCBP) must have a negative urine pregnancy test within 24 hours preceding receipt of first and second vaccine doses.
* WOCBP must use medically acceptable contraception.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.

Exclusion Criteria:

* Previously received an H5N1 influenza vaccine or who plan to receive an H5N1 influenza vaccine while participating in the study
* An acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses
* Medications or treatments that may adversely affect the immune system
* An active neoplastic disease or a history of any hematological malignancy. For this criterion, "active" is defined as having received treatment within the past 5 years.
* A long-term use of supraphysiologic doses of oral or parenteral steroids, or high-dose inhaled steroids within the preceding 6 months.
* A history of documented autoimmune disease.
* Pregnant, nursing mothers or women planning a pregnancy between enrollment and 42 days after randomization
* Prior serious reaction to any influenza vaccine
* History of Guillain-Barré Syndrome
* History of anaphylactic-type reaction to injected vaccines
* History of illicit drug use or alcohol abuse in the year preceding the study
* Received a seasonal influenza vaccine six months prior to enrollment
* Received any licensed inactivated or recombinant vaccine within 2 weeks prior to enrollment or any licensed live vaccine within 1 month prior to enrollment.
* Acute illness or fever within three days prior to study enrollment
* Participating in a study that involves an experimental agent or have received an experimental agent within 1 month prior to enrollment in this study, or who expect to receive another experimental agent during participation, or intend to donate blood during the 42-day primary study period.
* Received or expect to receive immunoglobulin or another blood product within the 3 months prior to enrollment in this study.
* An elevated liver function enzyme of ALT at baseline, regardless of the appraisal of clinical significance.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 341 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Treanor, MD, Principal Investigator — University of Rochester
Locations (5):
- United States (5):
  - Meridian Clinical Research, Omaha, Nebraska
  - University of Rochester Center for Vaccine Studies, Rochester, New York
  - Benchmark Reseach, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Treanor JJ, Chu L, Essink B, Muse D, El Sahly HM, Izikson R, Goldenthal KL, Patriarca P, Dunkle LM. Stable emulsion (SE) alone is an effective adjuvant for a recombinant, baculovirus-expressed H5 influenza vaccine in healthy adults: A Phase 2 trial. Vaccine. 2017 Feb 7;35(6):923-928. doi: 10.1016/j.vaccine.2016.12.053. Epub 2017 Jan 11. PMID 28089141
- See also: sponsor — http://www.proteinsciences.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PanBlok 15µg in 2% SE | PanBlok 3.8µg in 2% SE | PanBlok 7.5µg No Adjuvant | PanBlok 7.5µg in 2% SE
Started | 84 | 86 | 85 | 86
Completed | 75 | 81 | 78 | 76
Not Completed | 9 | 5 | 7 | 10
Not completed — Lost to Follow-up | 6 | 4 | 4 | 8
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Healthy adults 18-49 years of age with no prior vaccination with H5 pandemic influenza
Groups:
- Total: Total of all reporting groups
Arm/Group | PanBlok 15µg in 2% SE | PanBlok 3.8µg in 2% SE | PanBlok 7.5µg No Adjuvant | PanBlok 7.5µg in 2% SE | Total
Number analyzed (Participants) | 84 | 86 | 85 | 86 | 341
Age, Continuous [Mean (Full Range); unit: years] | 32 [19 to 48] | 31 [18 to 49] | 32 [18 to 49] | 30 [18 to 49] | 31 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 58 | 49 | 48 | 207
  Male | 32 | 28 | 36 | 38 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 1 | 4
  Asian | 2 | 3 | 1 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 3 | 0 | 7
  Black or African American | 28 | 22 | 21 | 25 | 96
  White | 52 | 58 | 56 | 58 | 224
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 12 | 12 | 42
  Not Hispanic or Latino | 76 | 76 | 73 | 74 | 299
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 84 | 86 | 85 | 86 | 341

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Seroconversion/Immunogenicity Between rHA Formulated in an oil-in- Water Adjuvant (SE) Compared to a rHA Antigen Alone.
Description: Immunogenicity was assessed by measuring the percentage of subjects in each group exhibiting seroconversion on Day 42. The treatment groups that received adjuvanted rHA were evaluated against a non-adjuvanted rHA treatment group for whether they demonstrated seroconversion rates and 95% confidence intervals.
Time Frame: 42 Days
Population: All subjects who received both doses of study vaccine and had pre- and post-immunization immunogenicity data for the time period summarized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PanBlok 15µg in 2% SE | PanBlok 3.8µg in 2% SE | PanBlok 7.5µg No Adjuvant | PanBlok 7.5µg in 2% SE
Number analyzed (Participants) | 76 | 81 | 80 | 76
percentage of participants | 83 [72.5 to 90.6] | 70 [59.2 to 80] | 9 [3.6 to 17.2] | 76 [65.2 to 85.3]

2. Secondary Outcome: Reactogenicity Immediately After Each Injection, Extending to Day 7.
Description: Solicited events of local and systemic reactogenicity Days 0-7. These events are expected to occur and not considered or recorded as Adverse Events.
Time Frame: 7 Days
Population: All randomized subjects who received at least one dose of study vaccine and provided any safety data following vaccination.
Measure: Number; unit: participants
Arm/Group | PanBlok 15µg in 2% SE | PanBlok 3.8µg in 2% SE | PanBlok 7.5µg No Adjuvant | PanBlok 7.5µg in 2% SE
Number analyzed (Participants) | 82 | 86 | 84 | 84
participants
  Elevated temperature | 0 | 0 | 0 | 0
  Fatigue | 6 | 9 | 9 | 9
  Chills | 3 | 0 | 2 | 3
  Arthralgia | 4 | 2 | 4 | 4
  Myalgia | 11 | 17 | 7 | 13
  Headache | 8 | 19 | 13 | 8
  Nausea/Vomiting | 1 | 6 | 8 | 3
  Diarrhea | 4 | 4 | 7 | 3
  Injection site pain | 34 | 34 | 6 | 32
  Injection site tenderness | 47 | 52 | 8 | 46
  Injection site erythema | 0 | 1 | 1 | 2

3. Secondary Outcome: Long-term Safety
Description: Incidence of Serious Adverse Events (SAEs), New Onset of Chronic Illnesses (NOCIs) and Adverse Events of Special Interest (AESIs) over 12 months following vaccination. Study subjects were followed every three months (for one year following Day 42) by telephone and visit for reports of SAEs, NOCIs, and AESIs.
Time Frame: 13 Months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | PanBlok 15µg in 2% SE | PanBlok 3.8µg in 2% SE | PanBlok 7.5µg No Adjuvant | PanBlok 7.5µg in 2% SE
Number analyzed (Participants) | 84 | 86 | 85 | 86
participants
  SAEs | 0 | 2 | 1 | 2
  NOCIs | 0 | 0 | 0 | 0
  AESIs | 0 | 0 | 0 | 0

4. Primary Outcome: The Difference in Geometric Mean Titer Between rHA Formulated in an oil-in- Water Adjuvant (SE) Compared to a rHA Antigen Alone.
Time Frame: 42 Days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | PanBlok 15µg in 2% SE | PanBlok 3.8µg in 2% SE | PanBlok 7.5µg No Adjuvant | PanBlok 7.5µg in 2% SE
Number analyzed (Participants) | 76 | 81 | 80 | 76
titer | 121.7 [88.2 to 168] | 76.1 [53.2 to 108.8] | 7.1 [5.9 to 8.4] | 77.5 [56 to 107.2]

ADVERSE EVENTS:
Time Frame: All AEs collected Days 0-42; Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) and New Onset Chronic Illnesses (NOCIs) collected through month 13 following vaccination.
Arm/Group | PanBlok 15µg in 2% SE | PanBlok 3.8µg in 2% SE | PanBlok 7.5µg No Adjuvant | PanBlok 7.5µg in 2% SE
Serious Adverse Events (participants affected / at risk) | 0/84 | 2/86 | 1/85 | 2/86
Other Adverse Events (participants affected / at risk) | 22/84 | 13/86 | 24/85 | 16/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PanBlok 15µg in 2% SE (N=84) | PanBlok 3.8µg in 2% SE (N=86) | PanBlok 7.5µg No Adjuvant (N=85) | PanBlok 7.5µg in 2% SE (N=86)
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 — History of clinical depression since adolescence
Community-acquired pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 — pneumonia complicated by pleural effusion
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Complicated by dehydration
Small bowel obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — History of abdominal surgery in childhood; irritable bowel syndrome
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PanBlok 15µg in 2% SE (N=84) | PanBlok 3.8µg in 2% SE (N=86) | PanBlok 7.5µg No Adjuvant (N=85) | PanBlok 7.5µg in 2% SE (N=86)
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 3 | 1
Fatigue (General disorders) | 3 | 1 | 3 | 0
Pain (General disorders) | 1 | 0 | 3 | 0
Fungal infection (Infections and infestations) | 0 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 1 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 1 | 2 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 4 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less